CLINICAL TRIAL: NCT05404919
Title: Utilization of Hepatitis B Virus Nucleic Acid Test Positive Donors for Hepatitis B Vaccinated Lung Transplant Candidates
Brief Title: Utilization of Hepatitis B Virus NAT+ Donors for Hepatitis B Vaccinated Lung Transplant Candidates
Acronym: INHIBITOR
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient enrollment; departure of primary investigator from institution
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Andrew M Courtwright, Assistant Professor of Medicine, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 851257
Record Dates: First submitted 2022-05-07; First posted 2022-06-03 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Lung Transplant; Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — hepatitis B hyperimmune globulin; entecavir; Tenofovir; tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Recipient of Hepatitis B NAT+ Donor (Other): All subjects will then be treated with Hepatitis B Immune Globulin and entecavir, tenofovir disoproxil, or tenofovir alafenamide (choice of specific drug to be based on long-term cost, clinical response, and renal function)
  Interventions: Drug: Hepatitis B Immune Globulin and entecavir, tenofovir disoproxil, or tenofovir alafenamide

INTERVENTIONS:
Drug: Hepatitis B Immune Globulin and entecavir, tenofovir disoproxil, or tenofovir alafenamide — Anti-hepatitis B medications

SUMMARY:
The objective of this study is to determine the safety and efficacy of transplanting lungs from hepatitis B virus (HBV) nucleic acid test positive (NAT+) donors into HBV vaccinated HBV surface antibody positive (sAb+) lung transplant candidates, who will then be treated with Hepatitis B Immune Globulin (HBIG) and entecavir, tenofovir disoproxil, or tenofovir alafenamide.

DETAILED DESCRIPTION:
Despite advances in organ preservation and the use of increasingly sophisticated bridge-to-transplant therapies, there is significant waitlist mortality among lung transplant candidates. Between 2017-2019, 637 patients died while awaiting donor lungs and 403 became too sick for transplant. To increase the pool of available donors, many transplant programs in the United States now accept donors with active hepatitis C virus (HCV) infections. Transplant recipients are then treated with anti-viral therapy in the post-operative period.

Some kidney and lung transplant programs have extended this strategy to include donors with hepatitis B virus (HBV) viremia. Following transplant, recipients are treated with Hepatitis B Immune Globulin (HBIG) and life-long antiviral therapy. Published studies have shown decreased waitlist mortality among kidney recipients who receive HBV nucleic acid test positive (NAT+) organs without adverse impact on allograft or hepatic function. It is unknown, however, whether this can be a safe and effective strategy for lung transplant candidates.

The aim of this phase II clinical trial is to assess the safety and efficacy of accepting lungs from HBV NAT+ donors for HBV vaccinated lung transplant candidates. The study will enroll 10 subjects, who will be treated with HBIG and entecavir, tenofovir disoproxil, or tenofovir alafenamide following transplant. Outcomes will include rates of HBV viremia and time to undetectable viral level; rates of acute HBV-associated hepatitis and persistent HBsAg positivity at one year; and 1-year patient and graft survival.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Able to provide informed consent
* Willing and able to travel to the University of Pennsylvania for routine post-transplant study visits
* Pre-menopausal women must agree to use birth control in accordance with the Mycophenolate Risk Evaluation and Mitigation Strategy (REMS) following transplant
* Both men and women must agree to use at least one barrier method of birth control or remain abstinent following transplant due to risk of HBV transmission
* Appropriate HBV vaccine pre-transplant response, defined as HBV sAb ≥12.00 mIU/mL

Exclusion Criteria:

* Donor characteristics:

  * Donation after circulatory death donor
  * Hepatitis C Virus (HCV) NAT+
  * PaO2/FiO2 <300 on FiO2 = 100% and PEEP=5
  * Age >55 years
  * Smoking history >20 pack years
* Transplant candidate characteristics:

  * Age >70 years
  * Any chronic liver disease (excluding non-alcoholic fatty liver disease (NAFLD)) associated with persistently elevated liver enzymes
  * Significant fibrosis (≥F2 on Fibroscan or Fib4 ≥1.67 (for patients unable to complete Fibroscan and without liver disease risk factors))
  * Inadequate insurance coverage of entecavir, tenofovir disoproxil, or tenofovir alafenamide
  * Retransplant candidate
  * Current use of extracorporeal membrane oxygenation (ECMO) or mechanical ventilation as a bridge to lung transplantation
  * HIV infection
  * Chronic kidney disease with estimated glomerular filtrate rate less than 50 ml/min/1.73 m2
  * Small bowel dysmotility or plan for prolonged medications and/or nutrition via tube route in the post-transplant period
  * Significant human leukocyte antibody (HLA) sensitization (Calculated Panel Reactive Antibody (CPRA) ≥60%)
  * Planned or high likelihood of anti-thymocyte globulin induction immunosuppression or rituximab treatment
  * Known hypercoagulable states including positive antiphospholipid antibodies with prior venous or arterial thromboembolic events or Factor V Leiden or Prothrombin mutations with or without prior venous or arterial thromboembolic events
  * History of hypersensitivity or anaphylactic reaction to immune globulin or similar products
  * Receiving or anticipated to receive drugs with significant entecavir or tenofovir interactions including phenytoin/fosphenytoin, oxcarbazepine, phenobarbital, primidone, rifabutin, and rifampin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Rate of HBV viremia | 1 year
  HBV viremia rate in HBV vaccinated patients who receive a lung transplant from a HBV NAT+ donor.
Time to undetectable HV DNA | 1 year
  Time to undetectable HBV DNA rate in HBV vaccinated patients who receive a lung transplant from a HBV NAT+ donor.
Rate of acute HBV-associated hepatitis | 1 year
  Rates of acute HBV-associated hepatitis in HBV vaccinated patients who receive a lung transplant from a HBV NAT+ donor.
Rate of persistent HBV surface antigen positivity | 1 year
  Rates of persistent HBV surface antigen (HBsAg) positivity at one year in HBV vaccinated patients who receive a lung transplant from a HBV NAT+ donor.

SECONDARY OUTCOMES:
One year patient survival | 1 year
  One year patient survival among lung transplant patients who receive an organ from a HBV NAT+ donor.
One year graft survival | 1 year
  One year graft survival among lung transplant patients who receive an organ from a HBV NAT+ donor.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Courtwright, MD, PhD, Principal Investigator — Hospital of University of Pennsyvlania
Locations (1):
- Hospital of University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No